CLINICAL TRIAL: NCT04006613
Title: Effects of a Circuit Training on Balance Management in a State of Fatigue in Persons With Multiple Sclerosis
Brief Title: Effects of a Circuit Training on Balance in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIRCUIT_SM
Record Dates: First submitted 2019-05-29; First posted 2019-07-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Fatigue; Balance; Aerobic training
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circuit Training (Experimental): Structured intervention to improve aerobic capacity, balance and strength
  Interventions: Other: Circuit Training
- Usual Care (Active Comparator): Unstructured intervention to improve mobility and balance
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Circuit Training — 20 minutes of High Intensity Aerobic Training (HI) on treadmill: 2 minutes warm up + 4x 4 minutes HI+ 2 minutes of active recovery; 10 minutes of dynamic balance training; 10 minutes of functional strength training.
  Arms: Circuit Training
Other: Usual Care — Exercises aimed at improving mobility and balance
  Arms: Usual Care

SUMMARY:
The aim of the study is to evaluate the effects of a circuit training rehabilitation program on the perceived impact of fatigue in daily life situations and on gait and balance. Half of the participants will follow the circuit training program, while the other half will follow usual care rehabilitation programs.

DETAILED DESCRIPTION:
Approximately 80% of Persons with Multiple Sclerosis rates fatigue among the three most disabling symptoms. Aerobic, balance and strength training have already been proved effective in rehabilitation, especially for Persons with Multiple Sclerosis. Fifty-two Persons with Multiple Sclerosis will be randomly allocated to an experimental group or to a control group following usual care rehabilitation programs. Experimental group will follow a circuit training rehabilitation program which combines high intensity aerobic training with balance and strength training. The study aims to verify the effects of the circuit training program on fatigue and on balance in different contexts with respect to usual care rehabilitation programs and to investigate effects of rehabilitation on immunological markers.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of Multiple Sclerosis (Polman criteria);
* No relapses in the previous three months;
* Expanded Disability Status Scale < 6,5;
* Able to walk 20 meter with or without an assistive device;
* Able to stand for 30 second without aid;
* MiniMental State Examination >20;

Exclusion Criteria:

* Unable to understand the aim of the study or unable to sign the informed consent form;
* Subjects following a steroidal drug therapy or assuming drugs affecting cardiac function;
* Subjects with psychiatric disorders;
* Subjects with cardiovascular diseases for whom aerobic training is forbidden;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Modified Fatigue Impact Scale at 6-8 weeks | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Provides an assessment of the effects of fatigue in terms of physical, cognitive and psychosocial functioning. Participant rates on a 5 point Likert scale (from 0="never" to 4= "Almost Always") their agreement with 21 statements. Higher numbers indicate greater fatigue.

SECONDARY OUTCOMES:
Change from Baseline Modified Dynamic Gait Index at 6-8 weeks | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Assesses individual's ability to modify balance while walking during 8 specific tasks. Scoring system for each task is based on 3 aspects of walking performance: time to complete (min 0, max 3 points), gait pattern (min 0, max 3 points) and level of assistance (min 0, max 2 points). Total score ranges from 0 to 64 with greater scores indicating better performance.
Change from Baseline 6 Minutes Walking Test at 6-8 weeks | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Assesses distance walked over 6 minutes as a sub-maximal test of endurance capacity.
Change from Baseline 10 Meter Walking Test at 6-8 weeks | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Assesses walking speed over a short distance
Change from Baseline 5-Time-Sit-To-Stand at 6-8 weeks | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Is used to quantify functional lower limb strength. Time taken to stand up and sit down for 5 consecutive times.
Change from Baseline 12 item Multiple Sclerosis Walking Scale at 6-8 weeks | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Is a self report measure of the impact of MS on walking ability. The scoring gives a 1 (no limitation) to 5 (extreme limitation) option for each item.
Change from Baseline Hospital Anxiety and Depression Scale at 6-8 weeks | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  A two dimension scale to identify depression and anxiety. 14 items divided inti two 7 items subscales. The respondent rates each item on a 4 point scale (ranging from 0 to 3).Higher scores indicates greater anxiety and/or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Cattaneo, PhD, Study Director — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Fondazione Don Carlo Gnocchi Onlus, Milan, Italy